CLINICAL TRIAL: NCT04551092
Title: Neurofeedback-EEG-VR (NEVR) System for Non-opioid Pain Therapy
Brief Title: Neurofeedback-EEG-VR System for Non-opioid Pain Therapy
Acronym: NEVR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Period of performance expired
Sponsor: Quantum Applied Science & Research, Inc. (Industry)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R43DA050380 (NIH)
Record Dates: First submitted 2020-07-13; First posted 2020-09-16 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single (Experimental): Single group to receive intervention
  Interventions: Device: NEVR

INTERVENTIONS:
Device: NEVR — a non-invasive, non-pharmacological alternative to treat pain by combining an innovative electroencephalography (EEG)-based Neurofeedback solution in an immersive virtual reality (VR) environment.

SUMMARY:
This study will assess the feasibility of developing the Neurofeedback-EEG-VR (NEVR) system for non-opioid pain therapy. Subjects suffering from pain will undergo sessions involving VR and Neurofeedback training and their pain will be assessed.

DETAILED DESCRIPTION:
QUASAR and UCSD are conducting a clinical trial on 25 subjects to evaluate the feasibility of a novel Neurofeedback electroencephalography (EEG) Virtual Reality (VR) system aimed at reducing chronic pain. The NEVR device consists of a dry electrode EEG headset combined with a VR Head-Mounted Display (VR-HMD) device and neurofeedback software. This approach relies on retraining the brain's networks to reduce the perception of pain and does not involve pharmaceutical drugs. Patients with chronic lower back pain will be recruited by UCSD at its Altman Clinical & Translational Research Institute. Patients that meet the recruitment criteria will be asked to conduct 20 1-hour long sessions of EEG-based Neurofeedback in VR over the course of a couple of months. Pain assessment and device usability questionnaires will be conducted prior to and after the first and last sessions, and at intermediate time points. This will be a single arm clinical trial aimed at demonstrating the safety and viability of the NEVR device, with the primary outcome measure being the ability of patients to conduct all 20 sessions safely and comfortably. Secondary outcome measures include assessment of changes in pain perception, and of changes in EEG activity patterns.

ELIGIBILITY:
Inclusion Criteria:

* Chronic back pain that can be of multifactorial etiology inclusive of axial and radicular back pain
* Report a Numerical Rating Scale (NRS, or Visual Analog Score VAS) score of greater than 6/10
* Must be willing to for the duration of the study make no pharmacological adjustments or have additional Interventional therapies, as reported by the patient
* Must have the cognitive capacity to provide consent/assent
* Must be able to sit up in a chair during the recording session
* Must demonstrate understanding of the protocol, its purpose and subject participation
* Must be fluent in English

Exclusion Criteria:

* Measured head size too small or too large for the EEG equipment
* Any significant skull defect
* History of a recent craniotomy (within the last six months)
* Any signs of scalp inflammation, irritation, or abnormal skin conditions
* History of epilepsy or seizures
* Known allergies to any material to be used in this project
* Sight disabilities that make participation impractical
* Hair styles with thick braids or dread locks

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walid Soussou, PhD, Principal Investigator — Quantum Applied Science & Research (QUASAR), Inc.
Locations (1):
- Altman Clinical and Translational Research Institute, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Lead organization website — http://www.quasarusa.com
- See also: Subaward research site — https://actri.ucsd.edu/index.html
- See also: NIH Funding Initiative — http://heal.nih.gov

RESULTS

PARTICIPANT FLOW:
Groups:
- NEVR Study: Single group to receive intervention
  NEVR: a non-invasive, non-pharmacological alternative to treat pain by combining an innovative electroencephalography (EEG)-based Neurofeedback solution in an immersive virtual reality (VR) environment.
Period: Overall Study
Arm/Group | NEVR Study
Started | 11
Completed | 0
Not Completed | 11
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | NEVR Study
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data not collected about 5 subjects. Signed consent but contact was lost after that.
  Participants
    number analyzed (Participants) | 6
    Female | 5
    Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data not collected for 5 subjects. Subjects signed consent but follow up contact was unsuccessful.
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 5
    Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Completing the Study
Description: The researchers will calculate the percentage of patients who complete all 20 sessions of the study without any adverse effects nor any discomfort from the device or VR.
Time Frame: up to 6 months
Population: Shortly after recruitment commenced, the study site was shut down for COVID and when re-opened it was a vaccine test site. The vaccine tests received priority and the study was not able to be conducted before the project period ended. No subjects completed the protocol and thus analysis was not able to be conducted.
Measure: Count of Participants; unit: Participants
Arm/Group | NEVR Study
Number analyzed (Participants) | 11
Participants | 0

2. Primary Outcome: Patient Tolerance of Device
Description: The researchers will survey the subjects about their comfort of wearing the device after each session on a scale of 1-10, where 1 is intolerable, 5 is just tolerable, and 10 is most comfortable. The researchers refer to this as the Comfort Scale.
Time Frame: up to 6 months
Population: 4 subjects only completed 1 session and no further sessions were conducted. Each subject reported on the 1-10 Comfort Scale for 6 measures. Subjects were asked to rate comfort for each of the 6 items on a scale from 1-10, where 1 was intolerable, 5 was just tolerable and 10 most comfortable. Higher values indicate a better comfort rating for that item. The mean values indicate the mean of the subjects' scores, as the goal is to produce a comprehensive comfort score per subject on a 1-10 scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NEVR Study
Number analyzed (Participants) | 4
score on a scale
  Pressure Points | 3 (.71)
  Helmet Weight | 5.25 (1.48)
  Headset Tightness | 6 (1.41)
  Neck Muscle Tightness | 7.5 (1.66)
  Headache | 6.5 (1.5)
  Overall Comfort | 6.75 (1.3)

3. Primary Outcome: Adverse Effect on Pain
Description: Subjects' back pain will be assessed prior to and after the first, 10th and last sessions via the following standardized subjective, objective, behavioral and functional evaluation tests: 1) Numerical Rating Scale (NRS, or Visual Analog Pain Score (VAS), 2) The DALLAS scale; 3) Patient Assessment Global Change. The researchers will compare the before and after session results to determine if the sessions had a negative impact on the patients' perceived pain.
Time Frame: up to 6 months
Population: The assessments were not conducted prior to and after Session 1 for the 4 subjects who completed one session. The subject testing site was also a COVID treatment and vaccine testing site and the Subject Matter Expert was not available to conduct these assessments. There are no data for this measure.
Arm/Group | NEVR Study
Number analyzed (Participants) | 0

4. Secondary Outcome: Changes in Pain Perception
Description: The researchers will evaluate changes in pain perception over the course of the 20 sessions as determined by the pain questionnaires listed above. The researchers will plot the changes and calculate the percent change between the first to last measurement.
Time Frame: 6 months
Population: Only 4 subjects completed any sessions and each of these only completed one session. Thus it was not possible to plot a change from session to session. There are no data for this outcome.
Arm/Group | NEVR Study
Number analyzed (Participants) | 0

5. Secondary Outcome: Changes in EEG Activity Patterns
Description: The researchers will calculate synchrony in electroencephalographic (EEG) alpha band (at 10Hz) across the temporal and central electrodes over the course of the 20 sessions. The researchers will compare the percentage of synchrony changes inter- and intra-sessions.
Time Frame: up to 6 months
Population: No subjects completed the protocol. Only 4 subjects did one session each. The data from these subjects were not adequate to conduct this calculation and no further sessions were conducted in which to revise the collection methodology to ensure adequate collection. Comfort survey data were collected but EEG data were not properly saved by the researchers and thus were not usable.
Arm/Group | NEVR Study
Number analyzed (Participants) | 0

6. Secondary Outcome: Dose Response
Description: The researchers will analyze the relationship between the number of sessions completed and the reported pain score of each of the three pain scales, as well as the EEG alpha synchrony. The research team will calculate a trendline to determine if there is a positive or negative trend and calculate a correlation index.
Time Frame: up to 6 months
Population: No subjects completed the protocol. No subjects completed more than one session. Calculation not able to be conducted.
Arm/Group | NEVR Study
Number analyzed (Participants) | 0

7. Secondary Outcome: Signal Quality
Description: The researchers will also calculate the percentage of the acquired EEG signal that is deemed to be unusable due to contamination by noise or artifacts (other than EMG or blink artifacts), as defined by regions where the root mean square (RMS) signal amplitude exceeds 100 microV.
Time Frame: up to 6 months
Population: A researcher error in using the data collection software meant that EEG data for the 4 participants who did one session were not saved properly to be transmitted to QUASAR scientists for analysis. Training for the researcher was rectified once the issue was identified but no more sessions were conducted after that. There are no data for this outcome.
Arm/Group | NEVR Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | NEVR Study
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT04551092/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT04551092/ICF_001.pdf